CLINICAL TRIAL: NCT06688253
Title: Intravenous Human IgG1 Fc Fragment (Efgartigimod) in Myasthenic Crisis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: argenx (Industry)
Responsible Party: Principal Investigator, . Shahr Shelly MD, Specialist in Neurology and Immunology, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rambam271
Record Dates: First submitted 2024-11-05; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Myasthenia Gravis Crisis
Keywords: Myasthenia Gravis Crisis
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group with Efgartigimod (Experimental): Efgartigimod will be given to patients with MG CRISIS
  Interventions: Drug: IV efgartigimod
- Historical PLEX group (No Intervention): this group is the retrospective arm

INTERVENTIONS:
Drug: IV efgartigimod — IV efgartigimod
  Other Names: vyvgart
  Arms: Interventional group with Efgartigimod

SUMMARY:
Efgartigimod in Myasthenic Crisis Background Myasthenia gravis (MG) is a prevalent autoimmune disorder affecting neuromuscular junctions, characterized by weakness in skeletal muscles. It is associated with the production of autoantibodies, primarily targeting acetylcholine receptors (AchR), and is often complicated by myasthenic crisis, which can lead to severe respiratory failure. Current treatments primarily involve non-specific immunosuppression, which may not provide rapid relief.

Aim This study investigates the therapeutic impact of efgartigimod, an FcRn-targeting Fc fragment, on patients experiencing a myasthenic crisis. We hypothesize that efgartigimod is non-inferior to conventional treatments like intravenous immunoglobulin (IVIG) and plasma exchange (PLEX) in terms of clinical efficacy and safety.

Study Rationale Efgartigimod aims to reduce pathogenic IgG autoantibodies implicated in MG by accelerating their degradation. This targeted approach could provide faster symptom relief during acute exacerbations compared to existing therapies.

Objectives Primary Objective: To assess the non-inferiority of efgartigimod compared to PLEX and IVIG based on MG-ADL improvements.

Secondary Objectives: Evaluate safety, tolerability, length of hospital stay, respiratory parameters, need for additional therapies, and one-year outcomes.

Primary Endpoint MG-ADL Improvement: Defined as a ≥3-point improvement post-treatment. The comparison will be made using one-month post-treatment assessments, with follow-ups every three months.

Secondary Endpoints Safety and tolerability Length of hospital stay Changes in respiratory function Need for rescue therapy in case of clinical deterioration Sample Size The study will recruit 32 patients (16 historical group and 16 interventional group), calculated to detect significant differences in MG-ADL improvements with a significance level of 0.05 and power of 0.80.

Patient Recruitment Patients with a confirmed diagnosis of MG who present to the neurology department will be recruited and randomly assigned to either the efgartigimod treatment group or the historical control group receiving standard care (IVIG/PLEX).

Inclusion Criteria Adults > 18 years Confirmed MG diagnosis with generalized weakness (MGFA class II-V) Positive AchR or MuSK antibodies Evidence of myasthenic crisis Informed consent Exclusion Criteria Contraindications to efgartigimod Significant comorbidities affecting study participation Prior exposure to efgartigimod Ongoing infections or conditions exacerbating MG symptoms Recent major surgery or significant renal/hepatic dysfunction Planned Protocol Administer efgartigimod intravenously at 10 mg/kg weekly for four weeks. Total trial duration: 12 months for enrollment and treatment, followed by a 14-month follow-up.

DETAILED DESCRIPTION:
Study Rationale: The study rationale for investigating the effectiveness of IV efgartigimod in myasthenic crisis hinges on the need for treatments that can provide rapid and targeted relief from the acute exacerbations of MG, which are life-threatening. Current treatments, while potentially effective, can be associated with significant side effects and may not work swiftly enough to address the urgent needs of a myasthenic crisis. Efgartigimod, an FcRn antagonist, has been designed to reduce the circulating levels of pathogenic IgG autoantibodies, which are implicated in the pathophysiology of MG. By accelerating the degradation of these autoantibodies, efgartigimod could potentially offer a faster onset of action and improve clinical outcomes in patients during a myasthenic crisis

ELIGIBILITY:
Inclusion Criteria:

* -Age > 18
* MG diagnosis
* A confirmed diagnosis of Myasthenia Gravis (MG) with generalized muscle weakness, classified as MGFA class II, III, IVa, or IVb and V.
* Positive AchR or MuSK antibodies (max three patients of the total cohort) this will be tested in our center for all patients.
* Myasthenic crisis: Worsening of > 3 or an increase >1 MG-ADL points of a sub score of any individual MG-ADL item other than double vision or eyelid droop and its clinically significant by the investigator. Alternatively, weakness related to MG that is severe enough to necessitate intubation or delay Ex-tubation following surgery.
* Willingness to provide informed consent.

Exclusion Criteria:-Contraindications to Efgartigimod.

* Other significant medical conditions that may interfere with study participation.
* Prior exposure to Efgartigimod.
* Male patients who do not intend to use effective contraception during trail or within last dosing
* Pateints with worsening muscle weekness due to concurrent infection or medications known to exacerbate MG.
* Patients with known or active seropositive HBV,HCV, HIV.
* Patients with documented lack of clinical response to Flax.
* Use of any investigational drug within 3 month or 5 helf -lives prior to screening.
* Avidance of significant disease ,recent major surgery or renal/ hepatic function who can put patient at undue risk.
* Previous participation in clinic trail involving ARGX-113
* Vaccination recived whitin 4 weeks prior screening using live or attenuated vaccinations.
* Patient Calssified MGFA Class 1

  1. Pregnant and lactating women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
MG-ADL scores observed before and after treatment initiation | 14 month
  Descriptive statistics will be used to summarize the characteristics of the study population. Kaplan-Meier curves to estimate the probability of cancer over time in cumulative analysis curves. A two-tailed p-value <0.05 was considered statistically significant

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam- Department of Neurology, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No